CLINICAL TRIAL: NCT00183885
Title: A Phase II Study of Intra-arterial Chemotherapy With Cisplatin and Mitomycin-C
Brief Title: A Phase II Study of Intra-arterial Chemotherapy With Cisplatin and Mitomycin-C in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3L-03-1
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Mitomycin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cisplatin + Mitomycin-C (Experimental): CDDP 60mg/m2 + Mitomycin-C 12mg/m2
  Interventions: Drug: mitomycin-c, cisplatin

INTERVENTIONS:
Drug: mitomycin-c, cisplatin — Intra-arterial cisplatin 60 mg/m2 and mitomycin-C 12 mg/m2 every 8 weeks

SUMMARY:
This study is for people with cancer of the liver that cannot be completely removed by surgery. This study involves giving the drugs mitomycin-C and cisplatin, into an artery in the liver. Mitomycin-C is a drug that has been approved by the FDA to treat cancer of the stomach and pancreas. Mitomycin-C is a drug that causes cancer cells to die and prevents them from reproducing. Cisplatin is also a drug that has been approved by the FDA. Cisplatin is approved to treat cancer of the testes, ovaries, lung, esophagus, bladder, head and neck. Cisplatin is a drug that prevents cancer cells from reproducing. The purpose of this study is to see how long it takes subjects' tumor(s) to grow after receiving the study drugs. Another purpose of this study is to look at the side effects of this study therapy and how long subjects survive after receiving it.

An additional purpose of this study is to see how well we can predict subjects' response to the study therapy, based on blood and tumor tissue tests. These tests will measure the levels of genes (the cell's blueprint) in subjects' tumors and blood. These genes affect how people's bodies react to the cancer drugs.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable, histologically confirmed hepatocellular carcinoma with evident disease limited to liver.
* Tissue from tumor must be available. This may be paraffin embedded tissue from previous biopsy/resection or if it is not available, a repeat biopsy must be performed. The requirement for biopsy may be waived if alpha-fetoprotein is greater than 500 ng/mL and in the investigators opinion not explained by a concurrent hepatic inflammatory process.
* Patients must agree to have a 20 cc blood sample drawn in addition to routine labs with each cycle of chemotherapy.
* Patients must have measurable disease. If prior radiation therapy was administered, measurable disease must be outside the radiation field.
* Patients must have a Zubrod performance status of 0-2.
* Patients must have a predicted life expectancy of at least 12 weeks.
* Patients must have a pre-treatment granulocyte count (i.e., segmented neutrophils + bands) of greater than or equal to 1,500/mm3, a hemoglobin level of greater than or equal to 9 gm/dl, and platelet count greater than or equal to 50,000/mm3. The granulocyte requirement may be waived if in the investigator's opinion the lower count reflects hypersplenism with adequate bone marrow reserves.
* Patients must have adequate renal function as documented by a calculated creatinine clearance ≥ 60.
* Patients must have adequate hepatic function as documented by a serum bilirubin less than or equal to 2x the institutional upper limit of normal, regardless of whether patients have liver involvement secondary to tumor. Patients may not have ascites or the ascites must be responsive to diuretics.

Exclusion Criteria:

* Patients who have received prior chemotherapy for unresectable disease
* Patients with any active or uncontrolled infection, including known HIV infection. (Patients with active hepatitis B will be placed on lamivudine. Patients with active hepatitis C will be eligible if liver tests qualify (5.1.9)
* Patients with psychiatric disorders that would interfere with consent or follow-up. Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method.
* Patients with any other severe concurrent disease, which in the judgment of the investigator, would make the patient inappropriate for entry into this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2004-10-18 (Actual); Primary Completion 2013-05-28 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Syma Iqbal, M.D., Principal Investigator — U.S.C. / Norris Cancer Center
Locations (1):
- U.S.C. / Norris Comprehensive Cancer Center, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study opened in October 2004 and closed in February 2012. All subjects were seen and treated in the medical clinics at the University of Southern California.
Period: Overall Study
Arm/Group | Cisplatin + Mitomycin-C
Started | 76
Completed | 37
Not Completed | 39
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 6
Not completed — Withdrawal by Subject | 5
Not completed — Switched to alternative treatment | 8
Not completed — Treatment delayed too long | 4
Not completed — Developed second malignancy | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cisplatin + Mitomycin-C
Number analyzed (Participants) | 76
Age, Continuous [Mean (Full Range); unit: Years] | 61 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 44
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 23
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 18
  More than one race | 0
  Unknown or Not Reported | 29
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: A modified Response Evaluation Criteria In Solid Tumors (RECIST) will be used. The modification to RECIST is that although all lesions will be followed, only the treated lesions will be included in the assessment of response. Additionally, all lesions will be evaluated according to the following criteria: Presence of arterial enhancement: Yes or No. Complete Response (CR) = Absence of enhancing tumor areas, reflecting complete tissue necrosis. Partial Response (PR) = A decrease > 50% of enhanced areas, reflecting partial tissue necrosis. Stable Disease (SD) = A tumor response between PR and PD. Progression (PD) = An increase > 25% in the size of > 1 measurable lesion(s) or the appearance of new lesions in the treated area (ie, specific segment or lobe of liver targeted by the intra-arterial infusion).
Time Frame: Up to 2 years
Population: Patients with measurable tumor who complete one cycle, or who terminate treatment for reasons of toxicity, or who progress prior to completion of one cycle, will be included in analysis of tumor response.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin + Mitomycin-C
Number analyzed (Participants) | 76
Participants
  CR | 0
  PR | 7
  SD | 47
  PD | 11
  Inevaluable for Response | 11

2. Secondary Outcome: Number of Participants With Grade 3 or Higher Toxicity
Description: Toxicity will be assessed according to CTCAE version 3.0
Time Frame: Up to 1 year
Population: All eligible patients who begin treatment are included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Cisplatin + Mitomycin-C
Number analyzed (Participants) | 76
Participants | 75

ADVERSE EVENTS:
Time Frame: Up to 1 year
Description: Adverse events are assessed during regularly scheduled follow up.
Arm/Group | Cisplatin + Mitomycin-C
All-Cause Mortality (participants affected / at risk) | 44/76
Serious Adverse Events (participants affected / at risk) | 51/76
Other Adverse Events (participants affected / at risk) | 75/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin + Mitomycin-C (N=76)
Hemoglobin (Blood and lymphatic system disorders) | 3 (3)
Leukocytes (Blood and lymphatic system disorders) | 4 (6)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 19 (27)
Platelets (Blood and lymphatic system disorders) | 27 (48)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 9 (10)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 (1)
Anorexia (General disorders) | 5 (5)
Constipation (Gastrointestinal disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 3 (4)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Nausea (Gastrointestinal disorders) | 7 (10)
Vomiting (Gastrointestinal disorders) | 6 (6)
Esophageal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Liver dysfunction/failure (clinical) (Hepatobiliary disorders) | 1 (1)
Edema limb (General disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 8 (12)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Alkaline phosphatase increased (Investigations) | 1 (2)
Blood bilirubin increased (Investigations) | 5 (7)
Creatinine increased (Investigations) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 8 (8)
Pain (bladder) (Renal and urinary disorders) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cisplatin + Mitomycin-C (N=76)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (4)
Hemoglobin decreased (Blood and lymphatic system disorders) | 60 (119)
Leukocytes (total WBC) decreased (Blood and lymphatic system disorders) | 3 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 17 (47)
Platelets decreased (Blood and lymphatic system disorders) | 39 (96)
Hypertension (Cardiac disorders) | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 53 (97)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (Gastrointestinal disorders) | 6 (8)
Insomnia (General disorders) | 2 (3)
Weight loss (Investigations) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5)
Injection site reaction/extravasation changes (General disorders) | 6 (8)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3 (3)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 (4)
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 42 (66)
Ascites (non-malignant) (Gastrointestinal disorders) | 5 (6)
Constipation (Gastrointestinal disorders) | 6 (8)
Dehydration (Gastrointestinal disorders) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 14 (20)
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1 (1)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) (Oral cavity) (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 38 (59)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (19)
Hemorrhage, CNS (Nervous system disorders) | 1 (1)
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Skin and subcutaneous tissue disorders) | 2 (3)
Infection with normal ANC or Grade 1 or 2 neutrophils (Urinary tract NOS) (Infections and infestations) | 1 (1)
Infection with unknown ANC (Urinary tract NOS) (Infections and infestations) | 1 (1)
Edema: limb (General disorders) | 23 (37)
Edema: trunk/genital (General disorders) | 1 (1)
Edema: viscera (General disorders) | 1 (1)
ALT (SGPT) increased (Metabolism and nutrition disorders) | 33 (58) — ALT, SGPT (serum glutamic pyruvic transaminase)
AST (SGOT) increased (Metabolism and nutrition disorders) | 38 (65) — AST, SGOT(serum glutamic oxaloacetic transaminase)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 15 (22)
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 37 (59)
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 42 (70)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 2 (2)
Creatinine increased (Metabolism and nutrition disorders) | 7 (10)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 15 (23)
Lipase (Metabolism and nutrition disorders) | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 3 (4)
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4 (5)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 5 (5)
Confusion (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 17 (21)
Encephalopathy (Nervous system disorders) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1)
Mental status (Nervous system disorders) | 1 (1)
Mood alteration (Anxiety) (Nervous system disorders) | 3 (4)
Neuropathy: sensory (Nervous system disorders) | 3 (4)
Dry eye syndrome (Eye disorders) | 1 (2)
Vision-blurred vision (Eye disorders) | 1 (1)
Pain (Abdomen NOS) (Gastrointestinal disorders) | 23 (45)
Pain (Back) (Musculoskeletal and connective tissue disorders) | 2 (4)
Pain (Extremity-limb) (Musculoskeletal and connective tissue disorders) | 2 (3)
Pain (Head/headache) (Nervous system disorders) | 4 (4)
Pain (Joint) (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (Throat/pharynx/larynx) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain (General disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (9)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (12)
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cystitis (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Urinary frequency/urgency (Renal and urinary disorders) | 2 (3)
Urinary retention (including neurogenic bladder) (Renal and urinary disorders) | 1 (1)
Flu-like syndrome (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-10-01): https://cdn.clinicaltrials.gov/large-docs/85/NCT00183885/Prot_SAP_000.pdf